CLINICAL TRIAL: NCT03052192
Title: Biological Aging, Medication, Malnutrition and Inflammation Among Acutely Ill and Healthy Elderly.
Acronym: FAM-CPH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Clinical Research Centre (Unknown); Lundbeck Foundation (Other); Region Hovedstadens Apotek (Other Government)
Responsible Party: Principal Investigator, Ove Andersen, Head of Clinical Research Centre, Hvidovre University Hospital
Other Study IDs: FAM-CPH-cohort; H-16038786 (Other: Committees on Health Research Ethics); AHH-2016-067 (I-suite 04931) (Other: Danish Data Protection Agency)
Record Dates: First submitted 2017-01-05; First posted 2017-02-14 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Aging; Polypharmacy; Malnutrition; Inflammation; Emergency Service, Hospital
MeSH Terms: conditions — Malnutrition; Inflammation; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, buffy coat.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- FAM group (n=98): ≥65 years. Acutely admitted medical patients.
  Included consecutively at admission to the Acute Medical Department at Amager and Hvidovre Hospital and Rigshospitalet - Glostrup.
  Follow-up at 4 weeks and 56 weeks after discharge and at any readmissions in the study period.
  Participants are interviewed on physical, mental and nutritional status, tested for functional and cognitive status, and have anthropometry, biochemistry, blood pressure, and immune activity measured. Participants are followed in national registries for information on diagnoses, hospital admissions, health care services used, and mortality.
  If a patient uses ≥5 prescribed drugs before hospitalization, a medication review will be performed by a clinical pharmacist and a geriatrician.
  Sample size calculations were performed for each primary outcome, and the final sample size was based on the calculation for the eating validation scheme which resulted in the largest sample size.
- Control group 1 (n=54): ≥65 years. No hospital admissions within the past two years.
  Matched individually with patients in the FAM group by age, sex, and municipality.
  Examined at inclusion and 52 weeks after inclusion.
  Participants are interviewed on physical, mental and nutritional status, tested for functional and cognitive status, and have anthropometry, biochemistry, blood pressure, and immune activity measured. Participants are followed in national registries for information on diagnoses, hospital admissions, health care services used, and mortality.
- Control group 2 (n=60): 20-35 years No admissions due to chronic or critical illness within the past 5 years (except admissions related to child birth, abortion, appendicitis, poisoning, traumas, concussion etc.)
  Examined at inclusion and 4 weeks after inclusion. The examination includes a questionnaire about life style, a physical examination, and blood samples.

SUMMARY:
In this study, the investigators will investigate and characterize acute medical patients in order to optimize patient courses in the acute care departments, especially with regard to polypharmacy and undernourishment. In addition, the investigators will investigate underlying immunological mechanisms of chronic inflammation and biological aging in this population to improve the current knowledge and possibilities for preventing chronic diseases and acute hospitalization.

DETAILED DESCRIPTION:
Malnutrition:

Malnutrition among elderly is associated with frailty, including loss of weight, muscle mass, function and quality of life and also with an increased number of hospital admissions. In this study, the investigators aim to describe the development of and the risk factors for malnutrition from admission to 4 weeks after discharge, in addition the investigators wish to characterize the inflammatory state of the malnourished patients.

Inappropriate polypharmacy:

The broad variation among elderly in health, number of chronic diseases, organ function, biological age and function makes the prescription of drugs to this population a very complex task with a high risk of inappropriate medication. 5-30% of all non-elective admissions are caused by inappropriate medications, and many of these are preventable. Therefore, the investigators aim to investigate the feasibility of a pharmacist-geriatrician medication review in the acute care department and the effect on the Medication Appropriateness Index score (MAI-score) .

Chronic inflammation and biological aging:

Chronic inflammation and biological aging promote the development of age-related chronic diseases. There is a large variation in the rate of aging between individuals, in particular among the elderly. This means that the chronological age of a person often does not reflect its true state of aging, the biological age. This challenges the ability to provide appropriate care and to predict responses to treatment and interventions in elderly patients. The underlying causes and mechanisms of biological aging and chronic inflammation are not well understood. There are currently no validated methods for measuring biological age and no measures of chronic inflammation which can be used in an acute setting. Here, the investigators aim to test a novel model for chronic inflammation and investigate the role of the NLRP3 inflammasome, NFkB (nuclear factor kappa light chain enhancer of activated B cells) and miRNAs in biological aging and chronic inflammation.

The study is prospective with 3 groups of study participants: one group is included in the Acute Medical Department and two healthy control groups (one young and one older). The follow-up comprises two predefined examinations and any readmissions at our hospital. Furthermore, participants are followed in the national registries.

ELIGIBILITY:
FAM group:

Inclusion Criteria:

* ≥65 years
* Acute medical patient
* Understands and speaks Danish

Exclusion Criteria:

* Unable to cooperate cognitively
* Terminal patients
* Patients in isolation

Control group 1:

Inclusion Criteria:

* ≥65 years
* No hospital admissions within the past 2 years

Exclusion Criteria:

* Acute admissions within the past 2 years
* Auto-immune diseases
* Treatment with immunosuppressive or biological therapies

Control group 2:

Inclusion Criteria:

* 20-35 years
* Caucasian
* No admissions due to chronic or critical illness within the past 5 years (except admissions related to child birth, abortion, appendicitis, poisoning, traumas, concussion etc.)

Exclusion Criteria:

* Auto-immune or chronic diseases

Ages: 20 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three study groups; the FAM group, control group 1 and control group 2
Sampling Method: Probability Sample
Enrollment: 212 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Eating validation scheme score | From inclusion to 4 weeks after discharge
  Development in nutritional status and risk factors of malnutrition within the FAM group.
MAI score (Medication Appropriateness Index) | From inclusion to 4 weeks after discharge
  Difference in summed MAI-score per patient. MAI score between inclusion and first follow-up visit (FAM group)
NF-kB (Nuclear Factor Kappa light chain enhancer og activated B cells) activity | From inclusion to 56 weeks after discharge
  The development in NF-kB activity between the groups will be investigated. The association of NF-kB activity with biological ageing-measured by chronic inflammation, and loss of function and cognition-will also be investigated.
Chronic inflammation | From inclusion to 4 weeks after inclusion
  Stability and discriminative ability of new model for chronic inflammation (Control group 2)
NLRP3 activity | From inclusion to 56 weeks after discharge
  Difference in NLRP3 inflammasome activity between groups.

SECONDARY OUTCOMES:
Bodyweight (kg) | From inclusion to 4 and 56 weeks after discharge
  Development in bodyweight
Quality of life | From inclusion to 56 weeks after discharge
  EQ-5D-5L(EuroQol-5Dimentions-5Llevels), mini geriatric depression score
Medication under-prescribing | From inclusion to 4 weeks after discharge
  Assessment of underutilization Index (AOU)
Inflammation in malnourished patients | 4 weeks after discharge
  Characterize the level of inflammation in malnourished patients
Functional recovery score | From inclusion to 56 weeks after discharge
  Assessing activities of daily living to characterize development in physical performance
Cystatin C | From inclusion to 56 weeks after discharge
Cytokine concentrations | From inclusion to 56 weeks after discharge
  The concentration of cytokines at baseline and in response to stimulation will be measured
Cytometry | From inclusion to 56 weeks after discharge
  Characterization of immune cell subsets
miRNA | From inclusion to 56 weeks after discharge
  Levels of miRNA will be measured, and their association with NF-kB activity and biological ageing will be investigated.
NF-kB activation | From inclusion to 56 weeks after discharge
  The activation of NF-kB in response to stimulation.
C-reactive protein (inflammation) | From inclusion to 56 weeks after discharge
  Difference in inflammation between groups
Soluble urokinase plasminogen activator receptor (suPAR) (ng/ml) | From inclusion to 56 weeks after discharge
  The plasma level of suPAR is a measure of inflammation and can be used to assess the difference in inflammation between groups
Frequency of physicians' acceptance of suggested changes in medications | At inclusion and at 4 weeks after discharge in the FAM group

OTHER OUTCOMES:
Sit-to-stand test | From inclusion to 56 weeks after discharge
  Development in physical performance
Cognitive functional ability | From inclusion to 56 weeks after discharge
  Orientation memory concentration, mini mental state examination, Hopkins verbal learning test, trail making test, digit symbol substitution test
Waist circumference (cm) | From inclusion to 56 weeks after discharge
Handgrip strength (kg) of dominant hand | From inclusion to 56 weeks after discharge
  Development in physical performance
Habitual 4 m gait speed (m/s) | From inclusion to 56 weeks after discharge
  Development in physical performance
Plasma and serum concentrations of admission blood samples | From inclusion to 56 weeks after discharge
  Routinely analyzed physiological biomarkers measured in plasma and serum
Blood concentration of cholesterol and triglycerides | From inclusion to 56 weeks after discharge
Blood concentration of metabolic markers | From inclusion to 56 weeks after discharge
  Measurement of insulin, blood glucose, and HbA1c
Plasma concentration of active drug substances | From inclusion to 56 weeks after discharge
CMV-IgG (Cytomegalovirus-immunoglobulin G) | From inclusion to 56 weeks after discharge
  Cytomegalovirus IgG titer

CONTACTS AND LOCATIONS:
Overall Officials: Ove Andersen, MD, PhD, Study Chair — Hvidovre University Hospital; Morten B. Houlind, MSc, Principal Investigator — Hvidovre University Hospital; Juliette Tavenier, MSc, Principal Investigator — Hvidovre University Hospital; Line JH Rasmussen, MSc, Principal Investigator — Hvidovre University Hospital; Aino L Andersen, MSc, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Amager & Hvidovre Hospital, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bornaes O, Andersen AL, Houlind MB, Kallemose T, Tavenier J, Aharaz A, Nielsen RL, Jorgensen LM, Beck AM, Andersen O, Petersen J, Pedersen MM. Mild Cognitive Impairment Is Associated with Poorer Nutritional Status on Hospital Admission and after Discharge in Acutely Hospitalized Older Patients. Geriatrics (Basel). 2022 Sep 10;7(5):95. doi: 10.3390/geriatrics7050095. PMID 36136804